CLINICAL TRIAL: NCT00089479
Title: A Randomized, Open-label Study of the Effect of Adjuvant Therapy With Adriamycin Plus Cytoxan Followed by Taxotere or Taxotere Plus Xeloda on Overall Survival in Female Patients With High-risk Breast Cancer
Brief Title: A Study of Xeloda (Capecitabine) in Women With High-Risk Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO17629
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: capecitabine [Xeloda]; Drug: Taxotere
- 2 (Active Comparator)
  Interventions: Drug: Taxotere

INTERVENTIONS:
Drug: capecitabine [Xeloda] — 825mg/m2 po bid on days 1-14 of each 3 week cycle
  Arms: 1
Drug: Taxotere — 75mg/m2 iv on day 1 of each 3 week cycle
  Arms: 1
Drug: Taxotere — 100mg/m2 iv on day 1 of each 3 week cycle
  Arms: 2

SUMMARY:
This 2 arm study will compare the efficacy and safety of Taxotere + Xeloda, versus Taxotere alone, following a regimen of Adriamycin plus Cytoxan in women with high-risk breast cancer. Following 4 cycles of Adriamycin and Cytoxan, patients will be randomized to receive either 1)Taxotere 75mg/m2 iv on day 1 and Xeloda 825mg/m2 po bid on days 1-14 of each 3 week cycle or 2) Taxotere 100mg/m2 iv alone on day 1 of each 3 week cycle. The anticipated time on study treatment is until disease progression, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients 18-70 years of age;
* adenocarcinoma of the breast;
* previous invasive breast cancer if diagnosed >5 years before entering study;
* no evidence of metastatic disease.

Exclusion Criteria:

* history of severe hypersensitivity reaction to Taxotere;
* previous treatment with anthracycline, anthracenedione (mitoxantrone), or taxane;
* treatment with fluoropyrimidine (5-fluorouracil) within the last 5 years.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2611 (Actual)
Dates: Start 2002-08; Primary Completion 2010-06 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Houston, Texas, United States

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241

RESULTS

PARTICIPANT FLOW:
Groups:
- AC Then T: Adriamycin 60 mg/m^2 iv plus Cytoxan 600 mg/m^2 iv repeat every 3 weeks for 4 cycles followed by Taxotere 100 mg/m^2; repeat every 3 weeks for 4 cycles
- AC Then XT: Adriamycin 60 mg/m^2 iv plus Cytoxan 600 mg/m^2 iv repeat every 3 weeks for 4 cycles followed by Xeloda 825 mg/m^2 po (bid) [total daily dose is 1650 mg/m^2] Days 1-14 every 3 weeks for 4 cycles plus Taxotere 75 mg/m^2 iv every 3 weeks for 4 cycles
Period: Overall Study
Arm/Group | AC Then T | AC Then XT
Started | 1304 | 1307
Received Treatment | 1305 (Safety Population (includes 19 patients randomized to ACXT, who received ACT)) | 1283 (Safety Population (includes 5 patients randomized to ACT, who received ACXT))
Completed | 973 (total includes Completed and Alive in follow-up) | 1018 (total includes Completed and Alive in follow-up)
Not Completed | 331 | 289
Not completed — Death | 108 | 75
Not completed — Withdrawal by Subject | 86 | 107
Not completed — Lost to Follow-up | 137 | 107

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AC Then T | AC Then XT | Total
Number analyzed (Participants) | 1304 | 1307 | 2611
Age Continuous [Mean (Standard Deviation); unit: years] | 51.2 (8.81) | 50.6 (9.19) | 50.9 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1304 | 1307 | 2611
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival [Number of Events]
Description: Number of patients with/without recurrence of breast cancer, or death due to any cause.
Time Frame: Time from the date of randomization until the date of first event, or date last known to be event free if no event was reported. Patients were followed for an average of 5 years.
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
participants
  Patients with event | 164 | 140
  Patients without events | 1140 | 1167

2. Secondary Outcome: Overall Survival [Number of Events]
Description: Number of patients who died/were alive.
Time Frame: Time from the date of randomization to the date of death, or date last known to be alive. Patients were followed for an average of 5 years.
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
participants
  Patients with event | 108 | 75
  Patients without events | 1196 | 1232

3. Primary Outcome: Disease Free Survival [Time to Event]
Description: Disease free survival was measured as the time from the date of randomization until the date of first event (recurrence of breast cancer, or death due to any cause). Patients without event at the time of the analysis were censored using the date they were last known to be recurrent disease free.
Time Frame: as for outcome 1
Population: Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
months | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial. | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial.

4. Secondary Outcome: Overall Survival [Time to Event]
Description: Overall survival was measured as the time from the date of randomization to the date of death. Patients still alive at the time of the analysis were censored using the date they were last known to be alive.
Time Frame: as for outcome 2
Population: Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
months | NA [NA to NA] — The median time to death based on Kaplan-Meier estimates was not reached in this adjuvant trial due to low death rate. | NA [NA to NA] — The median time to death based on Kaplan-Meier estimates was not reached in this adjuvant trial due to low death rate.

5. Secondary Outcome: Breast Cancer Free Survival [Number of Events]
Description: Number of patients with/without recurrence of breast cancer, new primary breast cancer, or death related to the chemotherapy administered or due to breast cancer.
Time Frame: Time from the date of randomization to event, or date last known to be event free if no event was reported. Patients were followed for an average of 5 years .
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
participants
  Patients with event | 158 | 144
  Patients without events | 1146 | 1163

6. Secondary Outcome: Breast Cancer Free Survival [Time to Event]
Description: Breast cancer-free survival was measured as time from the date of randomization to the date of recurrence of breast cancer, new primary breast cancer, or death related to the chemotherapy administered or due to breast cancer. Patients without event at the time of the analysis were censored using the date they were last known to be recurrent disease free.
Time Frame: Time from the date of randomization to death, or date last known to be event free if no event was reported. Patients were followed for an average of 5 years.
Population: Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
months | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial. | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial.

7. Secondary Outcome: Disease Free Survival Including New Primary Breast Cancer as Event [Number of Events]
Description: Number of patients with/without recurrence of breast cancer, new primary breast cancer, or death due to any cause.
Time Frame: as for outcome 1
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
participants
  Patients with event | 169 | 154
  Patients without events | 1135 | 1153

8. Secondary Outcome: Disease Free Survival Including New Primary Breast Cancer as Event [Time to Event
Description: Time from the date of randomization until the date of first event (recurrence of breast cancer, new primary breast cancer, or death due to any cause). Patients without event at the time of the analysis were censored using the date they were last known to be recurrent disease free.
Time Frame: as for outcome 1
Population: Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
months | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial. | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial.

9. Secondary Outcome: Disease Free Survival Including Any New Cancer as Event [Number of Events]
Description: Number of patients with/without recurrence of breast cancer, any new cancer, or death due to any cause.
Time Frame: as for outcome 1
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
participants
  Patients with event | 200 | 177
  Patients without events | 1104 | 1130

10. Secondary Outcome: Disease Free Survival Including Any New Cancer as Event [Time to Event]
Description: Time from the date of randomization until the date of first event (recurrence of breast cancer, any new cancer, or death due to any cause). Patients without event at the time of the analysis were censored using the date they were last known to be recurrent disease free.
Time Frame: as for outcome 1
Population: Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AC Then T | AC Then XT
Number analyzed (Participants) | 1304 | 1307
months | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial. | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached in this adjuvant trial.

ADVERSE EVENTS:
Time Frame: Length of study
Description: Safety Analysis Population: Patients are assigned to treatment groups based on the treatment (T or XT) they received, patients who did not receive T or X were assigned to the treatment groups as randomized. AE summaries display AEs that occurred during the period 1st study treatment intake (AC) until 30 days after last study treatment intake.
Arm/Group | AC Then T | AC Then XT
Serious Adverse Events (participants affected / at risk) | 264/1305 | 200/1283
Other Adverse Events (participants affected / at risk) | 1301/1305 | 1283/1283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AC Then T (N=1305) | AC Then XT (N=1283)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 118 | 80
NEUTROPENIA (Blood and lymphatic system disorders) | 10 | 11
ANAEMIA (Blood and lymphatic system disorders) | 0 | 5
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
CELLULITIS (Infections and infestations) | 11 | 6
PNEUMONIA (Infections and infestations) | 10 | 4
SEPSIS (Infections and infestations) | 5 | 3
INFECTION (Infections and infestations) | 4 | 3
DEVICE RELATED INFECTION (Infections and infestations) | 4 | 1
NEUTROPENIC INFECTION (Infections and infestations) | 2 | 3
BREAST CELLULITIS (Infections and infestations) | 2 | 2
BREAST INFECTION (Infections and infestations) | 2 | 2
BRONCHITIS (Infections and infestations) | 2 | 2
NEUTROPENIC SEPSIS (Infections and infestations) | 2 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 1
WOUND INFECTION (Infections and infestations) | 1 | 2
BREAST ABSCESS (Infections and infestations) | 1 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 1
SINUSITIS (Infections and infestations) | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 0
ACUTE SINUSITIS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
DEVICE RELATED SEPSIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0
FEBRILE INFECTION (Infections and infestations) | 0 | 1
FUNGAL SKIN INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
HISTOPLASMOSIS (Infections and infestations) | 1 | 0
MASTITIS (Infections and infestations) | 1 | 0
MENINGITIS BACTERIAL (Infections and infestations) | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1
ORAL HERPES (Infections and infestations) | 1 | 0
OTITIS MEDIA (Infections and infestations) | 1 | 0
PAROTITIS (Infections and infestations) | 0 | 1
PERIDIVERTICULAR ABSCESS (Infections and infestations) | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 1
PLEURAL INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 1
SOFT TISSUE INFECTION (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
VOMITING (Gastrointestinal disorders) | 13 | 5
DIARRHOEA (Gastrointestinal disorders) | 10 | 4
NAUSEA (Gastrointestinal disorders) | 7 | 6
STOMATITIS ALL (Gastrointestinal disorders) | 4 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 2
COLITIS (Gastrointestinal disorders) | 3 | 2
CONSTIPATION (Gastrointestinal disorders) | 3 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
OESOPHAGITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
PYREXIA (General disorders) | 21 | 9
CHEST PAIN (General disorders) | 5 | 11
ASTHENIA (General disorders) | 2 | 2
FATIGUE (General disorders) | 2 | 1
HERNIA OBSTRUCTIVE (General disorders) | 1 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 1
THROMBOSIS IN DEVICE (General disorders) | 1 | 1
CATHETER SITE PAIN (General disorders) | 1 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0
DEVICE DISLOCATION (General disorders) | 1 | 0
MEDICAL DEVICE COMPLICATION (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1
PAIN (General disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 11 | 18
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 4 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 5
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 3
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 2
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 8 | 7
HYPOTENSION (Vascular disorders) | 2 | 3
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 2 | 0
THROMBOSIS (Vascular disorders) | 2 | 0
AORTITIS (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
VENOUS OCCLUSION (Vascular disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 5 | 3
CONVULSION (Nervous system disorders) | 1 | 3
HEADACHE (Nervous system disorders) | 2 | 2
MIGRAINE (Nervous system disorders) | 2 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
CARDIOMYOPATHY ACUTE (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
PALPITATIONS (Cardiac disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 | 0
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1
BREAST MASS (Reproductive system and breast disorders) | 1 | 0
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 1 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
VAGINAL LACERATION (Reproductive system and breast disorders) | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 1
RASH (Skin and subcutaneous tissue disorders) | 2 | 0
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
BREAST RECONSTRUCTION (Surgical and medical procedures) | 0 | 1
LYMPHADENECTOMY (Surgical and medical procedures) | 0 | 1
NEOPLASM PROPHYLAXIS (Surgical and medical procedures) | 1 | 0
PROPHYLAXIS (Surgical and medical procedures) | 1 | 0
SIMPLE MASTECTOMY (Surgical and medical procedures) | 1 | 0
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 1
ANXIETY (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 2
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1
BREAST PROSTHESIS USER (Social circumstances) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AC Then T (N=1305) | AC Then XT (N=1283)
NAUSEA (Gastrointestinal disorders) | 1125 | 1118
STOMATITIS ALL (Gastrointestinal disorders) | 848 | 980
DIARRHOEA (Gastrointestinal disorders) | 581 | 759
VOMITING (Gastrointestinal disorders) | 618 | 591
CONSTIPATION (Gastrointestinal disorders) | 552 | 596
DYSPEPSIA (Gastrointestinal disorders) | 289 | 389
ABDOMINAL PAIN (Gastrointestinal disorders) | 159 | 249
DRY MOUTH (Gastrointestinal disorders) | 82 | 146
DYSPHAGIA (Gastrointestinal disorders) | 65 | 133
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 94 | 86
HAEMORRHOIDS (Gastrointestinal disorders) | 91 | 87
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 64 | 101
ORAL PAIN (Gastrointestinal disorders) | 65 | 87
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 42 | 69
FLATULENCE (Gastrointestinal disorders) | 31 | 70
ALOPECIA (Skin and subcutaneous tissue disorders) | 1113 | 1069
PALMAR-PLANTAR (Skin and subcutaneous tissue disorders) | 232 | 779
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 433 | 491
RASH (Skin and subcutaneous tissue disorders) | 357 | 316
DRY SKIN (Skin and subcutaneous tissue disorders) | 125 | 177
ERYTHEMA (Skin and subcutaneous tissue disorders) | 93 | 137
PRURITUS (Skin and subcutaneous tissue disorders) | 88 | 98
FATIGUE (General disorders) | 1123 | 1157
PYREXIA (General disorders) | 369 | 339
OEDEMA PERIPHERAL (General disorders) | 324 | 305
ASTHENIA (General disorders) | 196 | 179
OEDEMA (General disorders) | 184 | 139
CHILLS (General disorders) | 147 | 165
PAIN (General disorders) | 114 | 116
CHEST PAIN (General disorders) | 83 | 89
NEUTROPENIA (Blood and lymphatic system disorders) | 966 | 964
ANAEMIA (Blood and lymphatic system disorders) | 729 | 667
LEUKOPENIA (Blood and lymphatic system disorders) | 491 | 443
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 87 | 66
DYSGEUSIA (Nervous system disorders) | 450 | 534
HEADACHE (Nervous system disorders) | 413 | 464
NEUROPATHY PERIPHERAL (Nervous system disorders) | 327 | 259
DIZZINESS (Nervous system disorders) | 205 | 258
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 227 | 187
PARAESTHESIA (Nervous system disorders) | 109 | 99
HYPOAESTHESIA (Nervous system disorders) | 68 | 50
MYALGIA (Musculoskeletal and connective tissue disorders) | 671 | 566
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 616 | 503
BONE PAIN (Musculoskeletal and connective tissue disorders) | 218 | 177
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 186 | 187
BACK PAIN (Musculoskeletal and connective tissue disorders) | 166 | 152
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 69 | 61
COUGH (Respiratory, thoracic and mediastinal disorders) | 295 | 302
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 222 | 258
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 246 | 214
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 89 | 146
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 113 | 97
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 61 | 78
DECREASED APPETITE (Metabolism and nutrition disorders) | 440 | 455
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 306 | 278
DEHYDRATION (Metabolism and nutrition disorders) | 131 | 110
HYPOKALAEMIA (Metabolism and nutrition disorders) | 68 | 75
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 165 | 159
CANDIDIASIS (Infections and infestations) | 112 | 134
SINUSITIS (Infections and infestations) | 106 | 103
URINARY TRACT INFECTION (Infections and infestations) | 106 | 98
PHARYNGITIS (Infections and infestations) | 70 | 119
ORAL CANDIDIASIS (Infections and infestations) | 84 | 84
RHINITIS (Infections and infestations) | 66 | 78
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 75 | 56
INSOMNIA (Psychiatric disorders) | 381 | 397
DEPRESSION (Psychiatric disorders) | 218 | 182
ANXIETY (Psychiatric disorders) | 214 | 183
NEUTROPHIL COUNT DECREASED (Investigations) | 132 | 118
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 117 | 116
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 101 | 123
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 83 | 104
HAEMOGLOBIN DECREASED (Investigations) | 93 | 85
WEIGHT DECREASED (Investigations) | 67 | 50
HOT FLUSH (Vascular disorders) | 373 | 347
FLUSHING (Vascular disorders) | 114 | 158
LYMPHOEDEMA (Vascular disorders) | 124 | 71
LACRIMATION INCREASED (Eye disorders) | 452 | 396
VISION BLURRED (Eye disorders) | 74 | 95
EAR PAIN (Ear and labyrinth disorders) | 65 | 69
DYSURIA (Renal and urinary disorders) | 77 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.